CLINICAL TRIAL: NCT06517355
Title: Acceptability and Benefits of an Onco-sexology Program for Laryngectomy Patients and Their Partners
Acronym: ABSENS
Status: Recruiting | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 24 VADS 01
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: ORL Cancer
Keywords: ORL cancer; Onco-sexology care; Laryngectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with cancer (ORL) treated by laryngectomy
  Interventions: Other: In this research, the procedure under study is represented:

INTERVENTIONS:
Other: In this research, the procedure under study is represented: — * On the one hand, by carrying out sexology consultations which consist of individual interviews with a qualified sexologist nurse.
  * Secondly, questionnaires to assess quality of life and sexual function, to be completed by patients during standard follow-up consultations; and a questionnaire on satisfaction with sexological follow-up, to be completed by patients and their partners (if applicable) during the last standard follow-up consultation.

SUMMARY:
Single-centre prospective pilot study designed to demonstrate the acceptability of onco-sexology management for laryngectomy patients and their partners in order to improve their perception of their intimate life. This is a non-interventional study (category 3 Loi Jardé), which will not result in any change in patient management. All procedures will be carried out in accordance with standard practice.

Patients will be followed for 14 months.

ELIGIBILITY:
Inclusion Criteria:

For patients:

1. Patient to be treated for ORL cancer by total (pharyngo)laryngectomy
2. Patient WHO 0-1-2
3. Age greater than or equal to 18 years
4. Patient who has not objected to participation in the study.

For partners (if applicable) :

1. Age greater than or equal to 18 years
2. Subject who has not objected to participation in the study.

Exclusion Criteria:

For patients:

1. Patient with another co-existing malignant disease at the time of inclusion.
2. Any psychological, familial, geographical or sociological condition that does not allow for compliance with the medical follow-up and/or procedures foreseen in the study protocol.
3. Patients deprived of their liberty or under legal protection (guardianship and tutorship, safeguard of justice).

For partners (if applicable):

1. Patients deprived of their liberty or under legal protection (guardianship and tutorship, safeguard of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer (ORL) treated by laryngectomy.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is defined as the rate of patients meeting the acceptability criteria for onco-sexology management. | 14 months for each patient
  This rate corresponds to the ratio of the number of patients meeting the acceptability criteria to the total number of patients included.
  Acceptability is defined when the following two criteria are validated:
  * Completion of onco-sexology consultations 2 and 3 (at 3 and 12 months after cancer treatment)
  * Patient satisfaction ≥ 3 on a numerical scale from 1 to 5.

SECONDARY OUTCOMES:
For the patients: Patients' sexual satisfaction will be assessed using the specific scale of the EORTC QLQSHQ-C22 questionnaire. | 14 months for each patient
  The score, which ranges from 0 to 100, is determined according to the algorithm published by the EORTC, based on answers to 8 questions. This is a self-administered questionnaire validated in French
For the patients: Quality of life will be assessed using the EORTC QLQ-C30 questionnaire and the disease-specific QLQ-H&N43 questionnaire. | 14 months for each patient
  These are self-administered questionnaires validated in French.
For the patients: The female sexual function (desire, arousal, pain, lubrication, satisfaction, orgasm). | 14 months for each patient
  The FSFI (Female Sexual Function Index) is a self-administered questionnaire validated in French. It comprises 19 items studying 6 dimensions of female sexual function (desire, arousal, pain, lubrication, satisfaction, orgasm) which make up an overall score of between 2 and 36.
For the patients: The ability to have sexual intercourse by considering several domains (erections, ejaculations, desire and satisfaction). | 14 months for each patient
  The MSHQ (Male Sexual Health Questionnaire) is a self-questionnaire validated in French which assesses the ability to have sexual intercourse by considering several domains (erections, ejaculations, desire and satisfaction).
For the patients: The impact of (pharyngo)laryngectomy totale on the couple's relationship. | 14 months for each patient
  It will be assessed using a descriptive analysis (marital status before and after cancer treatment, stability, strengthening or deterioration of the couple's relationship).
For the patients: Satisfaction or dissatisfaction with the onco-sexology consultation. | 14 months for each patient
  It will be assessed using a Likert scale. This type of scale was developed to measure attitudes and opinions (Rensis Likert 'A Technique for the Measurement of Attitudes', Archives of Psychology, vol.140, 1932, p. 1-55).
For the partner: - The rate of partners verifying the acceptability criteria for onco-sexology management is defined by the ratio of the number of partners verifying the acceptability criteria to the total number of partners included. | 14 months for each partner
  The definition of acceptability is the same as for the primary endpoint.
For the partner: The impact of the (pharyngo)laryngectomy totale on the couple's relationship will be assessed using a descriptive analysis (stability, reinforcement or deterioration of the couple's life). | 14 months for each partner
For the partner: Satisfaction or dissatisfaction with the onco-sexology consultation will be assessed using a Likert scale. | 14 months for each partner

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France